CLINICAL TRIAL: NCT02221089
Title: Effect of Retaron® on Oxygen Induced Retinal Vasoconstriction in LPS Induced Inflammatory Model in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, assoc. Prof. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-090911
Record Dates: First submitted 2013-01-31; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Imparied Retinal Vascular Reactivity; Healthy Subjects
Keywords: Effect of Retaron on imparied retinal vascular reactivity after LPS administration in healthy subjects
MeSH Terms: interventions — endotoxin, Escherichia coli; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Retaron (Experimental)
  Interventions: Drug: Escherichia coli Endotoxin; Dietary Supplement: Retaron®
- Placebo (Placebo Comparator)
  Interventions: Drug: Escherichia coli Endotoxin; Other: Placebo

INTERVENTIONS:
Drug: Escherichia coli Endotoxin — dose: 2 ng/kg bodyweight (corresponding to 20 IU/kg), i.v. bolus on both study days.
  Other Names: LPS, US Standard Reference Endotoxin
Dietary Supplement: Retaron® — Dosage 1 capsule Retaron® per day.: Lutein 10mg, Zeaxanthin 2mg, Fishoil 500mg (with 250 mg DHA, 30 mg EPA), Vitamin C 100mg, Zinc 10mg, Selen 25µg, Vitamin E 25mg, Taurin 50mg, Aroniaextract 50mg, administered for 14 days
  Arms: Retaron
Other: Placebo — Placebo capsules identical in appearance to Retaron capsules
  Arms: Placebo

SUMMARY:
Oxidative stress has been implicated to play a pathogenic role in many disease processes, especially in age-related disorders such as age-related macular degeneration. It has been hypothesized that antioxidative agents such as vitamins and minerals, which are capable of scavenging free radicals, may reduce oxidative stress and may, in turn, be beneficial for patients with age-related disorders. Based on this hypothesis several different combinations of vitamins have been introduced, all targeting at reducing oxidative stress. However, the in-vivo effect of the antioxidative properties of a certain drug or vitamin combination is hard to investigate. In the current study, we propose to investigate the effect of Retaron®, a combination of carotoinoids, omega-3-fatty acids, a herbal extract of Aronia, vitamins and trace elements, in a systemic in-vivo inflammation model.

In the present study, the infusion of LPS, which is a cell wall component of gram-negative bacteria and a major mediator in the pathogenesis of septic shock, will be used as a standardized experimental model of systemic inflammation in humans. Given that inflammation is associated with enhanced oxidative stress and widespread endothelial dysfunction, the LPS model is well suitable for determination of the antioxidative effects of Retaron®. As a main outcome parameter the vascular reactivity of retinal vessels to systemic hyperoxia (induced by breathing 100% oxygen) will be tested in presence or absence of the antioxidant combination.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug, vitamins and minerals supplements as well
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Retinal Vascular Reactivity | Study day 1 and 2
  To investigate the effect of oral antioxidative supplementation (Retaron®) on impaired retinal vascular reactivity after LPS administration. Measurements will be performed using the Dynamic Vessel Analyzer (Imedos, Jena, Germany).

SECONDARY OUTCOMES:
Change in Ocular blood flow | Study day 1 and 2
  To investigate the effect of oral antioxidative supplementation on ocular blood flow during inflammation. Measurements will be performed using Laser Doppler Velocimetry (LDV) and the Blue Field entoptic technique.
Change in impaired endothelial function | Study day 1 and 2
  To investigate the effect of oral vitamins and minerals supplementation on impaired endothelial function caused by E. coli endotoxin as assessed by Laser Doppler Velocimetry, the Blue Field entoptic technique and the Dynamic Vessel Analyzer.
Change in antioxidative capacity | Study day 1 and 2
  To investigate the antioxidative capacity in the blood by determination of malondialdehyd (MDA) levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Kolodjaschna J, Berisha F, Lung S, Schaller G, Polska E, Jilma B, Wolzt M, Schmetterer L. LPS-induced microvascular leukocytosis can be assessed by blue-field entoptic phenomenon. Am J Physiol Heart Circ Physiol. 2004 Aug;287(2):H691-4. doi: 10.1152/ajpheart.01240.2003. Epub 2004 Mar 11. PMID 15016626
- [Background] Kolodjaschna J, Berisha F, Lasta M, Polska E, Fuchsjager-Mayrl G, Schmetterer L. Reactivity of retinal blood flow to 100% oxygen breathing after lipopolysaccharide administration in healthy subjects. Exp Eye Res. 2008 Aug;87(2):131-6. doi: 10.1016/j.exer.2008.05.006. Epub 2008 May 18. PMID 18614167
- [Background] Suffredini AF, Hochstein HD, McMahon FG. Dose-related inflammatory effects of intravenous endotoxin in humans: evaluation of a new clinical lot of Escherichia coli O:113 endotoxin. J Infect Dis. 1999 May;179(5):1278-82. doi: 10.1086/314717. PMID 10191237
- [Background] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Background] Violi F, Cangemi R. Antioxidants and cardiovascular disease. Curr Opin Investig Drugs. 2005 Sep;6(9):895-900. PMID 16187689